CLINICAL TRIAL: NCT00931515
Title: A Prospective, Multi-center, Randomized, Controlled Clinical Trial Evaluating the Safety and Effectiveness of NUBAC™ Disc Arthroplasty
Brief Title: Trial Evaluating the Safety and Effectiveness of NUBAC™ Disc Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pioneer Surgical Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N012009
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Degenerative Disc Disease
Keywords: DDD
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Total Disc Replacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NuBac (Experimental): NuBac device implanted at the L4/5 level
  Interventions: Device: NuBac
- Prodisc-L (Active Comparator): Prodisc-L implanted at the L4/5 level.
  Interventions: Device: Prodisc-L

INTERVENTIONS:
Device: NuBac — NuBac device implanted at the L4/5 level.
  Other Names: nucleus replacement; disc arthroplasty
  Arms: NuBac
Device: Prodisc-L — Prodisc-L implanted at the L4/5 level.
  Other Names: Total disc replacement
  Arms: Prodisc-L

SUMMARY:
The NuBac device is indicated for reconstruction following nucleotomy in skeletally mature patients at least 18 years of age with symptomatic single level degenerative disc disease (DDD) at L4/L5 only.

DDD is defined as discogenic back pain with or without leg pain; with degeneration of the disc as confirmed by patient history, physical examination, radiographic studies showing: decreased disc height, contained herniated nucleus, vacuum phenomenon (dark disc) OR positive discography at the affected level.

These DDD patients should have no more than Grade 1 spondylolisthesis at the involved level and should have failed at least six months of conservative, non-operative care.

Demonstrate non-inferiority compared to ProDisc.

DETAILED DESCRIPTION:
STUDY DESIGN:

Multicenter, prospective, randomized (1:1), controlled study comparing the artificial nucleus to ProDisc. After implanting artificial nucleus in two patients during the training session, enrollment of randomized patients shall begin. The study is expected to be completed in four years.

NUMBER OF INVESTIGATIONAL SITES and INVESTIGATORS:

10 - 20 investigational sites, 1 to 2 investigators per site, approximately 20-40 patients per site

ELIGIBILITY:
Inclusion Criteria:

* is at least 18 years of age and skeletally mature
* must have symptomatic single level degenerative disc disease at L4/5 requiring surgical treatment
* must have completed a minimum of six months of unsuccessful conservative, non-operative care
* must have discogenic back pain with or without leg pain
* must show radiographic confirmation using plain films, MRI, CT, myelogram or discography of one of the following: decreased disc height when compared to the adjacent level, contained herniated nucleus, or vacuum phenomenon (dark disc)
* must score at least 40% on the Oswestry Disability Index
* must score at least 4 on a 10cm Visual Analog Scale for back pain
* is able to comply with the protocol's follow-up schedule
* must understand and sign the informed consent document

Exclusion Criteria:

* symptomatic DDD at more than one level
* previous fusion at any lumbar level or laminectomy at the target level (discectomy, Intradiscal Electrothermal Annuloplasty, laminotomy, or nucleolysis performed > 6 months ago are permitted)
* clinically compromised vertebral bodies, at the affected level due to previous trauma, i.e., compression or burst fracture
* pars defect
* involved vertebral endplate dimensionally smaller than 34.5 mm in the medial-lateral direction and/or 27 mm in the anterior-posterior direction
* disc height less than 5 mm at the target level
* bony stenosis
* lytic spondylolisthesis, spondylolisthesis greater than 3mm
* lumbar scoliosis greater than 11 degrees.
* osteoporosis, osteopenia, osteomalacia, Paget's disease or metabolic bone disease
* Schmorl's nodes, an incomplete annulus, or endplates that are not intact
* spinal tumors
* symptomatic facet joint disease
* free fragment herniation confirmed radiographically
* isolated radicular compression syndrome, especially due to a disc herniation
* arachnoiditis
* active infection or surgical site infection
* is using any medication known to interfere with bone/soft tissue healing
* rheumatoid arthritis or other autoimmune disease
* systemic disease such as AIDS, HIV, hepatitis
* morbid obesity defined as body mass index (BMI) >40 or a weight more than 100 lbs over ideal body weight
* psychosocial disorders that would preclude accurate evaluation or has a history of substance abuse
* active malignancy except non-melanoma skin cancer; history of any invasive malignancy unless treated and in remission for at least five years
* documented allergies to metal or plastic; i.e., cobalt, chromium, molybdenum, polyethylene, titanium or polyetheretherketone
* pregnancy, or interested in becoming pregnant within the next two years
* prisoner
* involvement in an investigational drug or device study within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Songer, MD, Principal Investigator — Orthopedic Surgery Associates
Locations (17):
- United States (17):
  - Spine Group Beverly Hills, Beverly Hills, California
  - Tower Orthopedics & Sports Medicine, Beverly Hills, California
  - Bergey Spine Institute, Colton, California
  - Loma Linda University - Faculty Physicians, Loma Linda, California
  - University of Colorado, Anschutz Outpatient Pavilion, Aurora, Colorado
  - The Spine Institute, Loveland, Colorado
  - Florida Orthopaedic Institute, Tampa, Florida
  - Bone & Joint Physicians, Oak Lawn, Illinois
  - Heartland Hand & Spine Orthopedic Center, Merriam, Kansas
  - Orthopaedic Surgical Associates, Marquette, Michigan
  - The Orthopedic Center of St. Louis, St Louis, Missouri
  - Buffalo Neurosurgery, Buffalo, New York
  - Southern New York NeuroSurgical Group, Johnson City, New York
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - NeuroSpine Institute, Eugene, Oregon
  - Neurospine Solutions, PC, Bristol, Tennessee
  - Milwaukee Spinal Specialists, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from February 2009 to December 2010. Patients were recruited from the medical practices of the Investigators. Enrollment was stopped in December 2010 due to the slow enrollment rate. A total of 30 subjects participated in the study; the protocol was intended for 440 patients.
Pre-assignment Details: Two patients were enrolled in the study and received a patient identification number, but were never randomized to a treatment group and never implanted with the device. One patient decided not to participate prior to randomization. The second patient did not meet all inclusion/exclusion criteria.
Groups:
- NuBac: The NUBAC® disc arthroplasty system.
- ProDisc: The ProDisc® total disc replacement system.
Period: Overall Study
Arm/Group | NuBac | ProDisc
Started | 15 | 15
Completed | 13 | 10
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NuBac | ProDisc | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (11.2) | 40.1 (11.2) | 42.05 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 5 | 10 | 15
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Participants With Improved Patient Function
Description: The comparison of results was based on the proportion of participants with improved outcomes.
  The primary efficacy variable was treatment success based on the following criteria:
  1. Oswestry Disability Index score improved by at least 15 points
  2. Device success
  3. Neurological success
  4. Absence of major complications
  5. Absence of fusion at the index level A patient was considered a success upon meeting all five criteria. Failure to meet any of these criteria resulted in classification as a treatment failure.
Time Frame: 24 months
Measure: Number; unit: participants
Groups:
- ProDisc: The ProDisc® device total disc replacement system.
Arm/Group | NuBac | ProDisc
Number analyzed (Participants) | 13 | 10
participants | 7 | 6
Statistical Analysis 1: Comparison: NuBac vs ProDisc; Test type: Superiority or Other; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | NuBac | ProDisc
Serious Adverse Events (participants affected / at risk) | 3/15 | 0/15
Other Adverse Events (participants affected / at risk) | 11/15 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NuBac (N=15) | ProDisc (N=15)
Device expulsion (Surgical and medical procedures) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NuBac (N=15) | ProDisc (N=15)
Implant migration (Surgical and medical procedures) | 2 (2) | 0 (0)
Radiculitis (Nervous system disorders) | 0 (0) | 1 (1)
Back Pain (Nervous system disorders) | 5 (5) | 9 (9)
Hip/Buttock pain (Nervous system disorders) | 1 (1) | 3 (3)
Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leg paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Surgical site reaction (Surgical and medical procedures) | 0 (0) | 1 (1)
Adjacent level complication (Surgical and medical procedures) | 2 (2) | 4 (4)
Surgical treatment (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastrointestinal complication (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neck Cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Alopecia (General disorders) | 1 (1) | 0 (0)
Falling (General disorders) | 0 (0) | 1 (1)
Pregnancy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Psychiatric (Psychiatric disorders) | 0 (0) | 1 (1)
Shoulder Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Hand Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Because the study was stopped after a total of 30 patients, demonstration of non-inferiority was impossible. Results from the 2 groups were compared using the Fisher exact test for categorical variables and ANOVA for continuous variables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research parties agree not to make any publications of results until notified in writing by Sponsor that study is complete and results published in peer-reviewed journal; however if not published within 18 months, Research parties may pursue publication of individual results. Research parties must submit communication to Sponsor for review/approval at least 30 days prior to submission. Sponsor can require the modification of the manuscript or delay of publication.